CLINICAL TRIAL: NCT02710669
Title: Comparison of (R) and (S) Propafenone for Prevention of Atrial Fibrillation Induction
Brief Title: New Formulations of Propafenone to Treat Atrial Fibrillation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study halted/terminated prematurely due to COVID.
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bjorn Knollmann, Professor of Medicine and Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 151952; 1R01HL124935-01A1 (NIH)
Record Dates: First submitted 2016-03-12; First posted 2016-03-17 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Atrial Fibrillation
Keywords: ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Propafenone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- (R)-propafenone (Experimental): Single intravenous dose of (R)-propafenone (2mg/kg) infused over 10 minutes
  Interventions: Drug: (R)-propafenone
- (S)-Propafenone (Active Comparator): Single intravenous dose of (S)-propafenone (2mg/kg) infused over 10 minutes
  Interventions: Drug: (S)-Propafenone
- Placebo (Placebo Comparator): Placebo (normal saline) is infused over 10 minutes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: (R)-propafenone
  Arms: (R)-propafenone
Drug: (S)-Propafenone
  Arms: (S)-Propafenone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Propafenone is a currently used medicine to treat atrial fibrillation and is a mixture of two compounds, (R)-propafenone and (S)-propafenone. In this study, the investigators will randomize participants to (R)-propafenone, (S)-propafenone, or placebo.

DETAILED DESCRIPTION:
Atrial fibrillation is a common cardiac arrhythmia that needs development of more effective medications. Propafenone is a medicine currently used to treat atrial fibrillation and is a mixture of two compounds, (R)-propafenone and (S)-propafenone. The investigators have discovered that purified (R)-propafenone may be more effective than (S)-propafenone for treatment of atrial fibrillation, and that (S)-propafenone reduces the efficacy of (R)-propafenone when administered as a mixture. This study will compare the ability of (R)-propafenone, (S)-propafenone, and placebo to suppress the induction of atrial fibrillation in participants undergoing an atrial fibrillation ablation procedure.

ELIGIBILITY:
Inclusion:

1. History of atrial fibrillation
2. Greater than or equal to 18 years of age
3. Scheduled to undergo an atrial fibrillation ablation procedure
4. Able to provide written informed consent

Exclusion:

1. Long-standing persistent atrial fibrillation at the time of ablation (greater than 1 year of a continuous atrial fibrillation episode)
2. Is in atrial fibrillation or atrial flutter the morning of the ablation procedure
3. The presence of any of the following in a patient without a permanent pacemaker for implantable cardiac defibrillator

   1. sick sinus syndrome indicated by the inability to previously tolerate an antiarrhythmic drug due to bradycardia
   2. sinus bradycardia with a heart rate less than 50 beats per minute at the time of study drug administration
   3. right bundle branch block, left bundle branch block, or bifascicular block
   4. PR-interval > 280ms, or history of 2nd or 3rd degree atrioventricular block
4. Concomitant use of CYP3A4 and CYP2D6 inhibitors
5. Previous surgical or catheter ablation for atrial fibrillation or Cox-Maze procedure
6. Amiodarone use within 3 months prior to enrollment
7. Antiarrhythmic drug (other than amiodarone) within 5 half-lives prior to atrial fibrillation ablation
8. Expected life span < 1 year
9. Creatinine clearance <30 mL/min
10. Reversible cause of atrial fibrillation (ie. thyrotoxicosis)
11. Unrevascularized coronary artery disease
12. Canadian class IV angina
13. Left ventricular ejection fraction <40%
14. New York Heart Association Class III or IV symptoms
15. Previous heart transplantation
16. Planned heart transplantation or ventricular assist device
17. Cardiac/thoracic surgery <6 months prior to enrollment
18. Severe asthma or chronic obstructive pulmonary disease
19. Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2016-10; Primary Completion 2020-03-11 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Knollmann, MD/PhD, Principal Investigator — Vanderbilt University; Ben Shoemaker, MD, Study Director — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Faggioni M, Savio-Galimberti E, Venkataraman R, Hwang HS, Kannankeril PJ, Darbar D, Knollmann BC. Suppression of spontaneous ca elevations prevents atrial fibrillation in calsequestrin 2-null hearts. Circ Arrhythm Electrophysiol. 2014 Apr;7(2):313-20. doi: 10.1161/CIRCEP.113.000994. Epub 2014 Feb 3. PMID 24493699
- [Derived] Shoemaker MB, Yoneda ZT, Crawford DM, Akers WS, Richardson T, Montgomery JA, Phillips S, Shyr Y, Saavedra P, Estrada JC, Kanagasundram A, Shen ST, Michaud GF, Crossley G, Ellis CR, Knollmann BC. A Mechanistic Clinical Trial Using (R)- Versus (S)-Propafenone to Test RyR2 (Ryanodine Receptor) Inhibition for the Prevention of Atrial Fibrillation Induction. Circ Arrhythm Electrophysiol. 2022 Oct;15(10):e010713. doi: 10.1161/CIRCEP.121.010713. Epub 2022 Sep 27. PMID 36166682

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 193 participants were enrolled. 1 participant withdrew consent prior to randomization.
Groups:
- (R)-Propafenone: Single intravenous dose of (R)-propafenone (1mg/kg) infused over 10 minutes
  (R)-propafenone
- (S)-Propafenone: Single intravenous dose of (S)-propafenone (1mg/kg) infused over 10 minutes
  (S)-Propafenone
- Placebo: Placebo (normal saline) is infused over 10 minutes
  Placebo
Period: Overall Study
Arm/Group | (R)-Propafenone | (S)-Propafenone | Placebo
Started | 85 | 86 | 21
Completed | 71 | 75 | 19
Not Completed | 14 | 11 | 2
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Institutional delays (including COVID) | 2 | 2 | 0
Not completed — arrived in afib/aflutter | 10 | 8 | 2

BASELINE CHARACTERISTICS:
Population: One participant was not randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | (R)-Propafenone | (S)-Propafenone | Placebo | Total
Number analyzed (Participants) | 85 | 86 | 21 | 192
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [56 to 68] | 64 [57 to 70] | 59 [52 to 71] | 63 [56 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 35 | 8 | 81
  Male | 47 | 51 | 13 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 85 | 86 | 21 | 192
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3
  White | 84 | 83 | 20 | 187
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 85 | 86 | 21 | 192

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Induction of 30 Seconds of Atrial Fibrillation/Atrial Flutter
Description: A rapid atrial pacing protocol was used to attempt to induce atrial fibrillation/atrial flutter. Twenty minutes after start of the study drug, participants underwent placement of a decapolar coronary sinus catheter. Pacing was performed from the proximal electrode at 20 milliamps and a pulse width of 2 ms. Bursts from the CS proximal electrode were induced to attempt atrial fibrillation.
Time Frame: Twenty minutes post-dosage to end of induction protocol (approximately 10 minutes)
Population: 27 Participants not analyzed as follows: R GROUP: (1) prolonged pharmacy time compounding the study med; (8) arrived in atrial fib/flutter; (1) physician withdrew due to PAC's; (1) took antiarrhythmic prior to ablation; (1) difficult anatomy (1) ischemia on MRI; (1) Due to COVID the lab halted elective research. S GROUP: (7) arrived in afib; (1) clot on TEE; (1) elevated anxiety in patient; (1) procedure scheduled late in day; (1) cardiac cath work-up needed. PLACEBO GROUP: (2) arrived in afib
Measure: Count of Participants; unit: Participants
Arm/Group | (R)-Propafenone | (S)-Propafenone | Placebo
Number analyzed (Participants) | 71 | 75 | 19
Participants
  Sustained AF and/or AFL induced | 60 | 60 | 12
  Non-sustained AF and/or AFL induced | 11 | 15 | 7

2. Secondary Outcome: Number of Participants With Successful Inducibility of Atrial Fibrillation/Atrial Flutter Expressed as an Ordinal Variable Based on Stage of the Induction Protocol
Description: Inducibility of atrial fibrillation (AF) or atrial flutter (AFL) expressed as an ordinal variable based on stage of the induction protocol.
  * Stage 1 measured the AV block (Wenckebach) cycle length (AVBCL), AV node effective refractory period (AVN ERP) and atrial ERP (AERP). AVN ERP and AERP were measured at drive trains (S1) of 600 ms and 450 ms. Extrastimuli (S2) were introduced starting at a coupling interval of 500ms and decremented by 10ms with each pacing train.
  * Stage 2 consisted of 15-beat bursts from the CS proximal electrode. The starting cycle length was 250ms, which was decremented by 10ms with each burst. A 10-second rest period was used between bursts. Step 2 was complete when 1:1 atrial capture was lost or a minimum cycle length of 180ms was reached.
  Stage 3 consisted of 15-second bursts. The cycle length used for the bursts was the fastest cycle length achieved during Step 2 that maintained 1:1 atrial conduction.
Time Frame: Twenty minutes post-dosage to end of induction protocol (approximately 10 minutes)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | (R)-Propafenone | (S)-Propafenone | Placebo
Number analyzed (Participants) | 71 | 75 | 19
Participants
  Stage 1 | 5 | 5 | 1
  Stage 2 | 28 | 31 | 3
  Stage 3 | 27 | 24 | 8
  Non-inducible AF/AFL | 11 | 15 | 7

3. Secondary Outcome: Number of Participants With Successful Induction of 30 Seconds of Atrial Flutter
Description: A rapid atrial pacing protocol was used to attempt to induce atrial flutter. Twenty minutes after start of the study drug, participants underwent placement of a decapolar coronary sinus catheter. Pacing was performed from the proximal electrode at 20 milliamps and a pulse width of 2 ms. Bursts from the CS proximal electrode were induced to attempt atrial flutter.
Time Frame: Twenty minutes post-dosage to end of induction protocol (approximately 10 minutes)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | (R)-Propafenone | (S)-Propafenone | Placebo
Number analyzed (Participants) | 71 | 75 | 19
Participants
  Sustained AFL | 23 | 26 | 1
  Non-Sustained AFL | 48 | 49 | 18

ADVERSE EVENTS:
Time Frame: Adverse event information was collected the day of procedure only
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | (R)-Propafenone | (S)-Propafenone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/75 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/75 | 0/19
Other Adverse Events (participants affected / at risk) | 0/71 | 0/75 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT02710669/Prot_SAP_002.pdf
  • Informed Consent Form (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT02710669/ICF_001.pdf